CLINICAL TRIAL: NCT00765869
Title: A Randomised Controlled Trial of a Bowel Cancer Screening Decision Aid for Adults With Low Education and Literacy
Brief Title: Randomised Controlled Trial of a Literacy Sensitive Decision Aid for Bowel Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Dr Kirsten McCaffery, Screening and Test Evaluation program,University of Sydney
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HREC10403; ACTRN12608000011381
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Colorectal Neoplasms
Keywords: Decision support techniques
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Bowel cancer screening decision aid, DVD and Question Prompt List (QPL)
  Interventions: Other: Bowel cancer screening decision aid
- 2 (Experimental): Bowel cancer screening decision with DVD only
  Interventions: Other: Bowel cancer screening decision aid
- 3 (Active Comparator): Australian Government Bowel Cancer Screening consumer information booklet
  Interventions: Other: Australian Government Bowel Cancer Screening booklet

INTERVENTIONS:
Other: Bowel cancer screening decision aid — A decision aid developed for adults with low levels of education and literacy making decisions about bowel cancer screening, using faecal occult blood test (FOBT)
  Arms: 1
Other: Bowel cancer screening decision aid — A decision aid developed for adults with low levels of education and literacy making decisions about bowel cancer screening, using faecal occult blood test (FOBT)
  Arms: 2
Other: Australian Government Bowel Cancer Screening booklet — A consumer booklet developed by the Australian Government for people taking part in the National Bowel Cancer Screening program
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate a decision aid (written information booklet designed to facilitate informed decision making) to help people aged 55-64 years, with low levels of education and literacy, make an informed choice about bowel cancer screening, using faecal occult blood testing.

DETAILED DESCRIPTION:
Several countries have recently implemented national bowel cancer screening programs. To ensure equal access to screening, consumer information is needed to suit adults ranging in literacy level. Decision aids (DAs) are tools which have been developed to assist patients and consumers make informed health decisions and encourage active participation in health care decisions. Their use in a wide range of clinical settings has increased dramatically. However, most DAs are highly dependent upon high levels of literacy and numeracy, and few have been developed for low literacy populations.

This primary aims of this study are to assess the impact of the decision aid on (1) the proportion of adults who make an informed choice about bowel cancer screening (using faecal occult blood test) and, (2) the level of involvement in screening decisions among adults with lower levels of education and literacy.

There are three secondary aims of the study. First, to measure the effect of the decision support tool on decisional conflict, decision satisfaction, anxiety, and bowel cancer worry. Second, to identify participant's screening interest, intentions and behavior. Thirdly, we will explore participant's reactions towards the information materials they receive and whether the doctor influenced their screening decision.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 55-64 years
* Lower levels of education
* English as a main language spoken at home
* Average risk of bowel cancer

Exclusion Criteria:

* Higher levels of education
* Invitation to take part in bowel cancer screening in last two years
* Personal or strong family history of bowel cancer
* Had a bowel cancer screening test in the last two years

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 555 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-12 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Informed choice | 2 weeks post intervention
Involvement in screening decision | 2 weeks post intervention

SECONDARY OUTCOMES:
Anxiety | 2 weeks post intervention
Bowel cancer worry | 2 weeks post intervention
Decisional conflict | 2 weeks post intervention
Decision satisfaction | 2 weeks post intervention
Bowel cancer screening interest | 2 weeks post intervention
Bowel cancer screening intentions | 2 weeks post intervention
Screening behaviour | 2 weeks post intervention
Self reported bowel cancer symptoms | 2 weeks post intervention
Evaluation of intervention materials | 2 weeks post intervention
Influence of doctor on screening decision | 2 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: McCaffery J Kirsten, PhD, Principal Investigator — University of Sydney
Locations (1):
- Hunter Valley Research Foundation, Newcastle, New South Wales, Australia

REFERENCES:
- [Background] Smith SK, Trevena L, Nutbeam D, Barratt A, McCaffery KJ. Information needs and preferences of low and high literacy consumers for decisions about colorectal cancer screening: utilizing a linguistic model. Health Expect. 2008 Jun;11(2):123-36. doi: 10.1111/j.1369-7625.2008.00489.x. PMID 18494957
- [Derived] Stacey D, Lewis KB, Smith M, Carley M, Volk R, Douglas EE, Pacheco-Brousseau L, Finderup J, Gunderson J, Barry MJ, Bennett CL, Bravo P, Steffensen K, Gogovor A, Graham ID, Kelly SE, Legare F, Sondergaard H, Thomson R, Trenaman L, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2024 Jan 29;1(1):CD001431. doi: 10.1002/14651858.CD001431.pub6. PMID 38284415
- [Derived] Smith SK, Trevena L, Simpson JM, Barratt A, Nutbeam D, McCaffery KJ. A decision aid to support informed choices about bowel cancer screening among adults with low education: randomised controlled trial. BMJ. 2010 Oct 26;341:c5370. doi: 10.1136/bmj.c5370. PMID 20978060